CLINICAL TRIAL: NCT03823417
Title: The Effectiveness Of Intravenous Tranexamic Acid (TXA) on Reducing Perioperative Blood Loss For Patients Undergoing Periacetabular Osteotomy (PAO): A Randomized Double Blind Placebo Controlled Trial
Brief Title: The Effectiveness Of Intravenous TXA on Reducing Perioperative Blood Loss For Patients Undergoing PAO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigators decided not to begin the study.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Goobie, Associate Professor of Anaesthesiology, Harvard Medical School Associate in Perioperative Anesthesia, Boston Children's Hospital Clinical Director, Pharmacokinetics Laboratory., Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00030426
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Bleeding
Keywords: Tranexamic Acid; Periacetabular Osteotomy; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients who choose to participate will be randomized to receive either:
  1. placebo i.e. saline 0.9% (intravenous injection) (Control Group) or
  2. intravenous TXA given as a loading dose over 15 minutes of 30 mg/kg bolus (within an hour prior to surgical incision) and 10 mg/kg/hr infusion for the duration of the surgery
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal saline placebo (Placebo Comparator): the participant will get saline 0.9% intravenous infusion for the duration of the surgery
  Interventions: Drug: Normal saline
- Intravenous Tranexamic acid (Experimental): Intravenous TXA will be given as a loading dose over 15 minutes of 30 mg/kg bolus (within an hour prior to surgical incision) and 10 mg/kg/hr infusion for the duration of the surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous TXA given as a loading dose over 15 minutes of 30 mg/kg bolus (within an hour prior to surgical incision) and 10 mg/kg/hr infusion for the duration of the surgery
  Other Names: TXA
  Arms: Intravenous Tranexamic acid
Drug: Normal saline — Normal saline infusion
  Other Names: placebo
  Arms: Normal saline placebo

SUMMARY:
In this research study the investigators want to learn more about how a medication called tranexamic acid (TXA) could help reduce bleeding during Periacetabular Osteotomy (PAO) surgery. TXA is approved by the Food and Drug Administration (FDA) for the reduction of bleeding for many types of surgical procedures. TXA works by slowing the breakdown of blood clots and helps to prevent bleeding. From previous studies, TXA has been shown to effectively prevent bleeding in patients undergoing heart, spine and skull remodeling surgeries.

As PAO surgery has been associated with significant blood loss when compared to other types of joint surgeries. In order to try and avoid bleeding that may lead to complications, different strategies can be used. In this research study the investigators want to learn more about how a medication called tranexamic acid (TXA) could help reduce bleeding during PAO surgery.

DETAILED DESCRIPTION:
This prospective randomized placebo controlled double blind trial will enroll 80 adolescents and young adults undergoing elective peri-acetabular osteotomy (PAO). The primary aim is to determine if intravenous infusion of TXA during surgery is effective compared to standard care (no TXA) in decreasing blood loss (measured; and calculated) and blood transfusion (autologous and allogenic) perioperatively in adolescents and young adults presenting for PAO surgery. The rate of blood loss over time will be measured and compared between groups with adjustment for length of surgery (time; hours) and body weight (kg).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Age 13-35 years
* Scheduled for primary unilateral PAO +/- arthroscopy

Exclusion Criteria:

* Hematologic disorder, thrombocytopenia (Platelet count <140,000/uL3)
* Major hepatic, renal, or vascular disorder
* Active Thromboembolic disorder
* Color vision defect
* TXA allergy
* Taking anticoagulants or antiplatelet drugs (heparin, warfarin, clopidogrel)
* Ethical and/or religious objection to receiving blood products
* International patients
* Patients undergoing revision surgery
* Patients undergoing combined PAO and other surgeries such as surgical dislocation, proximal femoral osteotomy

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Blood loss | 1 week after surgery
  ml

SECONDARY OUTCOMES:
Plasma TXA level | 24 hours
  ug/mL

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goobie, MD, FRPCP, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston children hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maruyama M. CORR Insights((R)): Does Tranexamic Acid Reduce Blood Loss and Transfusion Requirements Associated With the Periacetabular Osteotomy? Clin Orthop Relat Res. 2015 Nov;473(11):3602-3. doi: 10.1007/s11999-015-4455-y. Epub 2015 Sep 9. No abstract available. PMID 26354175
- [Background] Sethna NF, Zurakowski D, Brustowicz RM, Bacsik J, Sullivan LJ, Shapiro F. Tranexamic acid reduces intraoperative blood loss in pediatric patients undergoing scoliosis surgery. Anesthesiology. 2005 Apr;102(4):727-32. doi: 10.1097/00000542-200504000-00006. PMID 15791100
- [Background] Goobie SM, Meier PM, Pereira LM, McGowan FX, Prescilla RP, Scharp LA, Rogers GF, Proctor MR, Meara JG, Soriano SG, Zurakowski D, Sethna NF. Efficacy of tranexamic acid in pediatric craniosynostosis surgery: a double-blind, placebo-controlled trial. Anesthesiology. 2011 Apr;114(4):862-71. doi: 10.1097/ALN.0b013e318210fd8f. PMID 21364458
- [Background] Wingerter SA, Keith AD, Schoenecker PL, Baca GR, Clohisy JC. Does Tranexamic Acid Reduce Blood Loss and Transfusion Requirements Associated With the Periacetabular Osteotomy? Clin Orthop Relat Res. 2015 Aug;473(8):2639-43. doi: 10.1007/s11999-015-4334-6. Epub 2015 May 20. PMID 25991434
- [Background] Goobie SM, Gallagher T, Gross I, Shander A. Society for the advancement of blood management administrative and clinical standards for patient blood management programs. 4th edition (pediatric version). Paediatr Anaesth. 2019 Mar;29(3):231-236. doi: 10.1111/pan.13574. PMID 30609198
- [Background] Goobie SM, Zurakowski D, Glotzbecker MP, McCann ME, Hedequist D, Brustowicz RM, Sethna NF, Karlin LI, Emans JB, Hresko MT. Tranexamic Acid Is Efficacious at Decreasing the Rate of Blood Loss in Adolescent Scoliosis Surgery: A Randomized Placebo-Controlled Trial. J Bone Joint Surg Am. 2018 Dec 5;100(23):2024-2032. doi: 10.2106/JBJS.18.00314. PMID 30516625
- [Background] Johnson DJ, Johnson CC, Goobie SM, Nami N, Wetzler JA, Sponseller PD, Frank SM. High-dose Versus Low-dose Tranexamic Acid to Reduce Transfusion Requirements in Pediatric Scoliosis Surgery. J Pediatr Orthop. 2017 Dec;37(8):e552-e557. doi: 10.1097/BPO.0000000000000820. PMID 29120963
- [Background] Goobie SM, Frank SM. Tranexamic Acid: What Is Known and Unknown, and Where Do We Go From Here? Anesthesiology. 2017 Sep;127(3):405-407. doi: 10.1097/ALN.0000000000001788. No abstract available. PMID 28696996